CLINICAL TRIAL: NCT05851053
Title: Breast Cancer Long-term Outcomes on Cardiac Functioning: a Longitudinal Study
Acronym: BLOC-II
Status: Recruiting | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor
Other Study IDs: 202100903
Record Dates: First submitted 2022-11-14; First posted 2023-05-09 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Neoplasm, Breast; Heart Failure; Cardiotoxicity; Ventricular Dysfunction
Keywords: Breast cancer; Cardiotoxicity; Heart failure
MeSH Terms: conditions — Breast Neoplasms; Heart Failure; Cardiotoxicity; Ventricular Dysfunction | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Breast cancer survivors: Survivors of BC, diagnosed ≥11 years ago, who received chemotherapy and/or radiotherapy
  Interventions: Diagnostic Test: Echocardiography
- Reference population: Age and GP matched reference population without a history of cancer
  Interventions: Diagnostic Test: Echocardiography

INTERVENTIONS:
Diagnostic Test: Echocardiography — During echocardiography, the following parameters will be assessed:
  * Dimensions
  * Left ventricle function
  * Right ventricle function
  * Valves: Aorta valve and pulmonic valve
  * Other findings such as: frequency, rhythm, quality

SUMMARY:
Rationale: In addition to surgery, effective breast cancer (BC) treatment typically requires chemotherapy, radiotherapy, or both. However, it is still unclear whether patients with BC are at increased risk of long-term cardiac dysfunction due to the adverse effects of these therapies. In a cross-sectional study in primary care, a comparison on cardiac dysfunction between 350 BC survivors and 350 age- and general practitioner (GP)- matched controls without cancer was made. In that study, BC survivors were at increased risk of mild systolic cardiac dysfunction (left ventricle ejection fraction (LVEF)< 54%). By contrast, there was no significant difference in an LVEF < 50% or in diastolic dysfunction. To date it remains uncertain whether the mild or subclinical dysfunction we observed predicts further cardiac deterioration. Consequently, the translation of these results into guidelines for the daily practice of the GP is unclear.

Objective: The aim of the here proposed study is to clarify whether cardiac function in survivors of BC should be monitored by GPs, by assessing whether an unselected population of long-term BC survivors is at increased risk of developing cardiac dysfunction, whether in this group at-risk subgroups exists, and what factors are associated with the highest risk.

Study design: A new assessment of cardiac function among women included in the BLOC-I study. This produces a longitudinal matched cohort design consisting of two cohorts in primary care.

Study population: Survivors of BC, diagnosed ≥11 years ago who received chemotherapy and/or radiotherapy, and a matched reference population with no history of cancer. All participants participated in the Breast cancer Long-term Outcome of Cardiac function (BLOC-I) study.

Main study parameters/endpoints: Left ventricular systolic dysfunction. Systolic cardiac dysfunction is defined as a LVEF <54/50/45%.

ELIGIBILITY:
Inclusion Criteria:

* Patients who previously took part in de BLOC-I study will be included. These criteria were:
* females diagnosed with stage I-III BC at least five years ago or local or locoregional recurrence of BC at least five years ago
* treatment with chemotherapy and/or radiotherapy.

Exclusion Criteria:

* Patients unfit to travel to the hospital due to severe mental or physical illness, based on assessment by their GP.

Exclusion criteria for the BC survivors in the BLOC-I study were:

* metastatic disease at the time of BC diagnosis;
* BC treatment after 80 years of age;
* history of treatment for other types of cancer.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: BC survivors were matched with women of the same age (±1 year) who had the same GP, but who had no history of cancer or cancer treatment (chemotherapy or radiotherapy).
  A longitudinal matched cohort design consisting of two cohorts in primary care: one with survivors of BC, diagnosed ≥11 years ago who received chemotherapy and/or radiotherapy, and one with a matched reference population with no history of cancer.
Sampling Method: Non-Probability Sample
Enrollment: 455 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Left ventricular systolic dysfunction | through study completion (from Ocotober 2022 - December 2024)
  Prevalance of systolic cardiac dysfunction defined as a LVEF <54%

SECONDARY OUTCOMES:
Clinically used LVEF cut-off points <45% and <50% | through study completion (from Ocotober 2022 - December 2024)
  Prevalance of systolic cardiac dysfunction defined as a LVEF <45% and <50%
Course of cardiac function | through study completion (from Ocotober 2022 - December 2024)
  Rate of change of systolic and diastolic cardiac function by change in LVEF
Cardiovascular diseases | through study completion (from Ocotober 2022 - December 2024)
  Prevalence of cardiovascular diseases obtained from electronic patient records
Symptoms of hearth failure | through study completion (from Ocotober 2022 - December 2024)
  Clinical symptoms of heart failure measured using a self-constructed questionnaire

OTHER OUTCOMES:
Patient characteristics | through study completion (from Ocotober 2022 - December 2024)
  age, BMI, menopausal state
Physical activity | through study completion (from Ocotober 2022 - December 2024)
  Changes in Physical Acticity measured with Short Questionnaire to Assess Health-enhancing physical activity (SQUASH)
Depression | through study completion (from Ocotober 2022 - December 2024)
  Symptoms of depression measured with Hospital Anxiety and Depression Scale - Despression (HADS-D)
Anxiety | through study completion (from Ocotober 2022 - December 2024)
  Symptoms of anxiety measured with Hospital Anxiety and Depression Scale - Anxiety (HADS-A)
Fatigue | through study completion (from Ocotober 2022 - December 2024)
  Multidimensional assessment of fatigue mesaured with Multidimensional Fatigue Index - 20 (MFI-20).
Use of cardiovascular medication | through study completion (from Ocotober 2022 - December 2024)
  Use of cardiovascular medication based on electronic patient records
Smoking behavior (self-reported pack years) | through study completion (from Ocotober 2022 - December 2024)
  Smoking behavior

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Boerman LM, Maass SWMC, van der Meer P, Gietema JA, Maduro JH, Hummel YM, Berger MY, de Bock GH, Berendsen AJ. Long-term outcome of cardiac function in a population-based cohort of breast cancer survivors: A cross-sectional study. Eur J Cancer. 2017 Aug;81:56-65. doi: 10.1016/j.ejca.2017.05.013. Epub 2017 Jun 8. PMID 28601706